CLINICAL TRIAL: NCT06207942
Title: Extended Follow-up Substudy of the Sedation, Temperature and Pressure After Cardiac Arrest and Resuscitation -STEPCARE Trial
Brief Title: Stepcare Extended Follow-up Substudy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); The George Institute for Global Health, Australia (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: extfustep2024
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Arrest With Successful Resuscitation; Hypoxia, Brain; Cognitive Impairment; Caregiver Burden
MeSH Terms: conditions — Hypoxia, Brain; Cognitive Dysfunction; Caregiver Burden | interventions — Deep Sedation

STUDY DESIGN:
Intervention Model Description: 2X2X2 factorial., with all participants taking part in each factor
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants (out of hospital cardiac arrest survivors and caregivers) will be blinded. Assessors of neurological prognosis will be blinded. Outcome assessors and investigators will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Sedation, temperature device and high MAP (Active Comparator)
  Interventions: Device: Feed back controlled temperature device; Other: High MAP; Other: Deep sedation
- Sedation, no temperature device and high MAP (Active Comparator)
  Interventions: Other: High MAP; Other: Deep sedation; Other: Fever control without a device
- Sedation, temperature device and low MAP (Active Comparator)
  Interventions: Device: Feed back controlled temperature device; Other: Deep sedation; Other: Low MAP
- Sedation, no temperature device, and low MAP (Active Comparator)
  Interventions: Other: Deep sedation; Other: Fever control without a device; Other: Low MAP
- Minimal sedation, temperature device, and high MAP (Active Comparator)
  Interventions: Device: Feed back controlled temperature device; Other: High MAP; Other: Minimal sedation
- Minimal sedation, no temperature device and high MAP (Active Comparator)
  Interventions: Other: High MAP; Other: Fever control without a device; Other: Minimal sedation
- Minimal sedation, temperature device and low MAP (Active Comparator)
  Interventions: Device: Feed back controlled temperature device; Other: Low MAP; Other: Minimal sedation
- Minimal sedation, no temperature device and low MAP (Active Comparator)
  Interventions: Other: Fever control without a device; Other: Low MAP; Other: Minimal sedation

INTERVENTIONS:
Device: Feed back controlled temperature device — If core temperature exceeds 37.7 degrees celsius a feedback controlled-device will be used at set to 37.5 degrees celsius
  Arms: Minimal sedation, temperature device and low MAP; Minimal sedation, temperature device, and high MAP; Sedation, temperature device and high MAP; Sedation, temperature device and low MAP
Other: High MAP — A mean arterial blood pressure (MAP) of >85mmHg will be used. Vasopressors will be titrated to this target during 36 hours
  Arms: Minimal sedation, no temperature device and high MAP; Minimal sedation, temperature device, and high MAP; Sedation, no temperature device and high MAP; Sedation, temperature device and high MAP
Other: Deep sedation — Deep sedation for at least 36 hours
  Arms: Sedation, no temperature device and high MAP; Sedation, no temperature device, and low MAP; Sedation, temperature device and high MAP; Sedation, temperature device and low MAP
Other: Fever control without a device — Management of fever in the intensive care unit without a device
  Arms: Minimal sedation, no temperature device and high MAP; Minimal sedation, no temperature device and low MAP; Sedation, no temperature device and high MAP; Sedation, no temperature device, and low MAP
Other: Low MAP — A mean arterial blood pressure (MAP) of >65mmHG will be used. Vasopressors will be titrated to this target during 36 hours
  Arms: Minimal sedation, no temperature device and low MAP; Minimal sedation, temperature device and low MAP; Sedation, no temperature device, and low MAP; Sedation, temperature device and low MAP
Other: Minimal sedation — A strategy of minimal sedation in the intensive care unit, used only as needed to facilitate transport, imaging and invasive procedures
  Arms: Minimal sedation, no temperature device and high MAP; Minimal sedation, no temperature device and low MAP; Minimal sedation, temperature device and low MAP; Minimal sedation, temperature device, and high MAP

SUMMARY:
To provide detailed information on long-term outcomes in relation to potential neuroprotection and improvements in recovery for different targets of sedation, temperature, and pressure management in post out of hospital cardiac arrest survivors at 6 and 12 months. In addition, the impact of caring for a post OHCA survivor will be explored.

DETAILED DESCRIPTION:
This extended follow-up substudy is incorporated into the multi-center, international, factorial randomized Sedation, Temperature and Pressure after Cardiac Arrest and Resuscitation -STEPCARE trial (Clinical trials identifier:NCT05564754) were out of hospital cardiac arrest participants will be randomized to different targets of sedation, temperature, and MAP management.

Only selected STEPCARE sites will participate in this extended follow-up substudy. At the extended follow up participating sites all out of hospital cardiac arrest participants randomized in the STEPCARE trial, who survive and provide consent, will be eligible to participate in this substudy, with no further inclusion or exclusion criteria.The extended follow-up substudy is estimated to enroll approximately 600 post OHCA survivors. One nominated caregiver per post OHCA survivor will be invited to be included in the study.

Participants will be followed up at 6 and 12 months.

The primary outcome for this extended follow up substudy is cognitive function at 6 months for the out of hospital cardiac arrest survivors andCaregiver burden at 6 months for the caregivers.

ELIGIBILITY:
All OHCA participants randomized in the STEPCARE trial at the extended follow-up participating sites, who survive and provide consent, with no further inclusion or exclusion criteria.

The inclusion and exclusion criteria for the STEPCARE trial are:

* Inclusion criteria: out-of-hospital cardiac arrest of non-traumatic origin, minimum of 20 minutes without chest compressions (defined as stable return of spontaneous circulation. ROSC), unconsciousness (defined as not being able to obey verbal commands equal to a FOUR-score motor response of <4, or being intubated and sedated because of agitation after sustained ROSC, eligible for intensive care without restrictions or limitation, inclusion within 4 hours (240 minutes) of ROSC (or 220 minutes of stable ROSC).
* Exclusion criteria: on ECMO prior to randomization, pregnancy, suspected or confirmed intracranial hemorrhage, previously randomized in the STEPCARE trial.

For caregivers, the eligibility will be that they live with, or have weekly or more frequent contact (in person or over the telephone) with the post OHCA survivor. Only one nominated caregiver per post OHCA survivor will be able to be included in the study. This would typically be the caregiver that would identify as the primary caregiver of the post OHCA survivor if needed, but may also be another close family member.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 6 months
  Cognitive function for out of hospital cardiac arrest survivors. Score range. Higher scores=better cognition
Zarit Burden Interview (ZBI) | 6 months
  Caregiver burden for caregivers to out of hospital cardiac arrest survivors. Score range 0-88. Higher scores= worse indicating more caregiver burden

OTHER OUTCOMES:
Symbol Digit Modalities Test (SDMT) | 6 and 12 months
  Processing speed. For out of hospital cardiac arrest survivors. Scores presented as age and education adjusted z-scores. Higher scores=better
Hospital Anxiety and Depression Scale (HADS) | 6 and 12 months
  Symptoms of anxiety and depression. For both out of hospital cardiac arrest survivors and caregivers. Score range 0-21 for anxiety and depression respectively. Higher scores=worse and incerased symptoms of anxiety and depression
Post Posttraumatic Stress Disorders Checklist updated for DSM-5 (PCL-5) | 6 and 12 months
  Symptoms of posttraumatic stress. For both out of hospital cardiac arrest survivors and caregivers. Score range 0-80. Higher scores=worse indicating increased symptoms of PTSD
Modified Fatigue Impact Scale (MFIS) | 6 and 12 months
  Impact of fatigue. For out of hospital cardiac arrest survivors. Score range 0-84. Higher scores= worse indicating more problems with impact of fatigue
modified Rankin Scale (mRS) | 12 months
  Functional outcome. For out of hospital cardiac arrest survivors. Score range 0-6. Higher scores= worse indicating a poorer functional outcome
World Health Organization Disability Assessment (WHODAS) 2.0 | 6 and 12 months
  Disability. For both out of hospital cardiac arrest survivors and caregivers. 36 item version score range 0-100. 12 item version score range 0-48. Higher scores=worse indicating more disability
Return to work | 6 and 12 months
  Questions about work prior to cardiac arrest and at time of follow up. For both out of hospital cardiac arrest survivors and caregivers. Categorical item
EuroQol health survey 5 dimensions 5 levels response version (EQ-5D-5L) | 12 months for out of hospital cardiac arrest survivors. 6 and 12 months for caregiver
  Health related quality of life. For both out of hospital cardiac arrest survivors and caregivers. For EQ dimensions score range 1-5 and higher scores=worse indicating more health problems. For EQ VAS score range is 0-100 with higher scores= better and representing higher satisfaction with overall health
Life satisfaction visual analogue scale from the World Value Survey | 6 and 12 months
  Life satisfaction. For both out of hospital cardiac arrest survivors and caregivers. Score range 1-10. Higher scores=better indicating better life satisfaction
Timed Stands Test (TST) | 6 and 12 months
  Lower extremity strength. For out of hospital cardiac arrest survivors. Raw score adjusted for gender and age and categorized as normal, problems or unable.
Jamar hand grip dynamometer | 6 and 12 months
  Upper extremity strength. For out of hospital cardiac arrest survivors. Raw scores age and gender adjusted and categorized as normal, problems or unable.

CONTACTS AND LOCATIONS:
Locations (34):
- Australia (8):
  - Princess Alexandra Hospital, Brisbane
  - The Sutherland Hospital, Caringbah
  - The Prince Charles Hospital, Chermside
  - Nepean hospital, Kingswood
  - St George hospital, Kogarah
  - Liverpool hospital, Liverpool
  - Austin hospital, Melbourne
  - Royal North Shore Hospital, Sydney
- Belgium (2):
  - Ziekenhuis Oost Limburg, Genk
  - Ghent university hospital, Ghent
- Finland (3):
  - Helsinki Helsingfors university central hospital, Helsinki
  - Jorvi hospital, Jorvi
  - Tampere university hospital, Tampere
- Germany (3):
  - Charite university hospital, Berlin
  - Universitäres Herzzentrum Lübeck Universitätsklinikum Schleswig-Holstein, Lübeck
  - Tubingen university hospital, Tübingen
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg
- New Zealand (4):
  - Auckland city hospital, Auckland
  - Middlemore hospital, Auckland
  - Christchurch hospital, Christchurch
  - Wellington hospital, Wellington
- Norway (2):
  - Sorlandet hospital, Arendal
  - Oslo university hospital Rikshospitalet, Oslo
- Sweden (5):
  - Sahlgrenska university hospital, Gothenburg
  - Hallands hospital, Hålland
  - Helsingborg hospital, Helsingborg
  - Skåne university hospital, Lund
  - Skåne university hopsital, Malmo
- Switzerland (2):
  - Bern university hospital, Bern
  - Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (4):
  - The Essex Cardiothoracic Centre, Basildon
  - Bristol Royal Infirmary, Bristol
  - University hospital of Wales, Cardiff
  - St Bartholomew's hospital, London

IPD SHARING:
Plan to Share IPD: Undecided
Upon resonable request following publication

REFERENCES:
- See also: Official STEPCARE trial website — https://stepcare.org/